CLINICAL TRIAL: NCT00433147
Title: A Randomized, Open-label Study to Assess the Safety and Tolerability of Multiple Dose Levels and Multiple Dosing Regimens of AT2101 in Adult Patients With Type 1 Gaucher Disease Currently Receiving Enzyme Replacement Therapy
Brief Title: A Study of AT2101 (Afegostat Tartrate) in Adult Patients With Type 1 Gaucher Disease Currently Receiving Enzyme Replacement Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GAU-CL-201
Record Dates: First submitted 2007-02-07; First posted 2007-02-09 (Estimated); Results first posted 2018-08-15 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-08

CONDITIONS: Gaucher Disease, Type 1; Type 1 Gaucher Disease; Gaucher Disease
Keywords: afegostat tartrate; isofagomine tartrate; AT2101; Amicus Therapeutics
MeSH Terms: conditions — Gaucher Disease | interventions — AT2101

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Afegostat tartrate 25 milligrams (mg) once per day (Experimental): Afegostat tartrate was administered orally during the 4-week treatment period.
  Interventions: Drug: Afegostat tartrate
- Afegostat tartrate 150 mg once per day (Experimental): Afegostat tartrate was administered orally once per day during the 4-week treatment period.
  Interventions: Drug: Afegostat tartrate
- Afegostat tartrate 150 mg once every four days (Experimental): Afegostat tartrate was administered orally once every 4 days during the 4-week treatment period.
  Interventions: Drug: Afegostat tartrate
- Afegostat tartrate 150 mg once every seven days (Experimental): Afegostat tartrate was administered orally once every 7 days during the 4-week treatment period.
  Interventions: Drug: Afegostat tartrate

INTERVENTIONS:
Drug: Afegostat tartrate
  Other Names: isofagomine tartrate; AT2101

SUMMARY:
This study was conducted to test the safety and tolerability of afegostat tartrate in participants with type 1 Gaucher disease already receiving enzyme replacement therapy.

DETAILED DESCRIPTION:
This was a Phase 2, open-label study in participants with Gaucher disease, a lysosomal storage disorder. Afegostat tartrate (also known as AT2101 or isofagomine tartrate) is designed to act as a pharmacological chaperone by selectively binding to misfolded β-glucocerebrosidase (GCase) and helping it fold correctly, intended to restore GCase activity. The study consisted of a 14-day screening period, a 28-day treatment period, and a 7-day wash-out period. Participants received 1 of 4 dosing regimens for afegostat tartrate.

ELIGIBILITY:
Inclusion Criteria:

* Had a confirmed diagnosis of type 1 Gaucher disease with a known documented missense gene mutation in at least 1 of the 2 gene-encoding β-glucosidase alleles
* Clinically stable
* Male or female participants, 18 to 74 years old inclusive
* All participants of childbearing potential used adequate birth control
* Provided written informed consent to participate in the study

Exclusion Criteria:

* Clinically significant disease, severe complications from Gaucher disease, or serious illness that precluded participation in the study in the opinion of the Investigator that compromised the safety of the participant or precluded the participant from completing the study
* During the screening period, any clinically significant findings, as deemed by the Investigator
* Partial or total splenectomy (removal of spleen) within the 2 years prior to study entry
* History of pulmonary hypertension or Gaucher related lung disease
* History of allergy or sensitivity to the study drug or any excipients, including any prior serious adverse reaction to iminosugars (for example, N-butyldeoxynojirimycin or miglustat)
* Pregnant or breast-feeding
* Current/recent drug or alcohol abuse
* Treatment with any investigational product in the 90 days before study entry
* Treatment in the previous 90 days with any drug known to have a well-defined potential for toxicity to a major organ
* Presence or symptoms of gastrointestinal, liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-03-23 (Actual); Primary Completion 2008-02-19 (Actual); Study Completion 2008-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Clinical Research, Study Director — Amicus Therapeutics
Locations (10):
- United States (10):
  - San Francisco, California
  - Coral Springs, Florida
  - Decatur, Georgia
  - Iowa City, Iowa
  - New York, New York
  - Cincinnati, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Houston, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were screened for evaluation of eligibility to participate in the study. Confirmatory β-glucosidase genotype testing was done at screening to confirm reported genotype. Thirty participants received at least 1 dose of study drug. All participants were eligible for inclusion in the safety and 29 in the pharmacodynamics (PD) populations.
Period: Overall Study
Arm/Group | Afegostat Tartrate 25 Milligrams (mg) Once Per Day | Afegostat Tartrate 150 mg Once Per Day | Afegostat Tartrate 150 mg Once Every Four Days | Afegostat Tartrate 150 mg Once Every Seven Days
Started | 7 | 7 | 9 | 7
Safety Population (All participants who received at least 1 dose of study drug.) | 7 | 7 | 9 | 7
PD Population (Participants in the Safety Population with a baseline and at least 1 post-baseline PD measurement.) | 7 | 6 | 9 | 7
Received at Least One Dose of Study Drug | 7 | 7 | 9 | 7
Completed | 7 | 6 | 9 | 7
Not Completed | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Afegostat Tartrate 25 mg Once Per Day: Afegostat tartrate was administered orally during the 4-week treatment period.
- Total: Total of all reporting groups
Arm/Group | Afegostat Tartrate 25 mg Once Per Day | Afegostat Tartrate 150 mg Once Per Day | Afegostat Tartrate 150 mg Once Every Four Days | Afegostat Tartrate 150 mg Once Every Seven Days | Total
Number analyzed (Participants) | 7 | 7 | 9 | 7 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (15.1) | 43.4 (18.0) | 36.7 (12.0) | 45.0 (12.3) | 41.3 (14.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 7 | 5 | 22
  Male | 2 | 2 | 2 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number Of Participants Who Experienced Severe Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were defined as any adverse event (AE) with a start date on or after administration of the study drug (on Day 1). A severe AE was defined as an AE that was incapacitating and required medical intervention. The number of participants who experienced 1 or more severe TEAEs after dosing on Day 1 through 7 days after the last dose of study drug (Day 35) is presented. A summary of serious and all other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Day 1 (after dosing) through Day 35
Population: Safety Population: all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Afegostat Tartrate 25 mg Once Per Day | Afegostat Tartrate 150 mg Once Per Day | Afegostat Tartrate 150 mg Once Every Four Days | Afegostat Tartrate 150 mg Once Every Seven Days
Number analyzed (Participants) | 7 | 7 | 9 | 7
Participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline To End Of Treatment In Beta-glucocerebrosidase (GCase) Levels In White Blood Cells (WBC)
Description: GCase is a biomarker used to assess the PD effects of afegostat tartrate. Blood samples were collected to assess GCase levels in WBC. The baseline value was defined as the last non-missing value before the start of study drug.
Time Frame: Baseline, Day 28
Population: PD Population: All participants who were included in the Safety Population and had a baseline and at least 1 post-baseline PD measurement.
Measure: Mean (Standard Deviation); unit: pmol/mg/min
Arm/Group | Afegostat Tartrate 25 mg Once Per Day | Afegostat Tartrate 150 mg Once Per Day | Afegostat Tartrate 150 mg Once Every Four Days | Afegostat Tartrate 150 mg Once Every Seven Days
Number analyzed (Participants) | 7 | 6 | 9 | 7
pmol/mg/min
  Baseline | 8.732 (3.1079) | 8.543 (4.1560) | 9.371 (3.5133) | 12.035 (5.4742)
  Day 28 | 19.148 (17.0210) | 23.557 (14.6970) | 14.687 (4.4901) | 13.026 (8.7286)
  Change from Baseline to Day 28 | 10.226 (16.4000) | 15.013 (11.2934) | 4.686 (3.1759) | -1.028 (3.8147)

ADVERSE EVENTS:
Time Frame: Day 1 (after dosing) to Day 35
Arm/Group | Afegostat Tartrate 25 mg Once Per Day | Afegostat Tartrate 150 mg Once Per Day | Afegostat Tartrate 150 mg Once Every Four Days | Afegostat Tartrate 150 mg Once Every Seven Days
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/9 | 0/7
Other Adverse Events (participants affected / at risk) | 4/7 | 2/7 | 4/9 | 1/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afegostat Tartrate 25 mg Once Per Day (N=7) | Afegostat Tartrate 150 mg Once Per Day (N=7) | Afegostat Tartrate 150 mg Once Every Four Days (N=9) | Afegostat Tartrate 150 mg Once Every Seven Days (N=7)
Dry eye (Eye disorders) | 0 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Platelets counts decreased (Investigations) | 1 | 0 | 1 | 0
Red blood cell count decreased (Investigations) | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Eyelids pruritus (Eye disorders) | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Sinus headache from seasonal allergies (General disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator can publish only the results from this trial, provided they supply the sponsor (or authorized entity) a copy of any proposed publication for review prior to submission for publication. If requested and prior to publication, the investigator will remove information deemed confidential or proprietary by the sponsor and will withhold publication for an additional period of time to allow the sponsor to take appropriate measures to establish and preserve its proprietary rights.